CLINICAL TRIAL: NCT00878917
Title: Randomized, Double-Masked, Active Controlled, Crossover Phase III Equivalence Study of Dorzolamide 2% Eye Drops Solution In Subjects With Open Angle Glaucoma Or Ocular Hypertension
Brief Title: Equivalence Study of Dorzolamide 2% Eye Drops Solution
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alfred E. Tiefenbacher (GmbH & Co. KG) (Industry)
Responsible Party: Dr. Harm Peters, Alfred E. Tiefenbacher (GmbH & Co. KG)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DOR/2008
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Equivalence Study; Eye Drops Solution; Dorzolamide; Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — dorzolamide; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dorzolamide (Experimental)
  Interventions: Drug: Dorzolamide 2 % eye drops solution

INTERVENTIONS:
Drug: Dorzolamide 2 % eye drops solution — 1 drop into eye(s) three times a day for the duration of each treatment phase

SUMMARY:
The study aims to prospectively prove the equivalence of the test product and the reference solution in lowering intraocular pressure in patients with open angle glaucoma and ocular hypertension. For this purpose the patients are randomized into two sequences of study drug administration in a crossover study with an adequate wash-out period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of any race aged 18 years or older
* A clinical diagnosis of open angle glaucoma, pseudoexfoliation or pigment dispersion glaucoma, or ocular hypertension in one or both eyes
* IOP controllable on one drug treatment in the study eye in way that assures clinical stability of vision and the optic nerve throughout the study
* Baseline IOP between 18 and 32 mmHg in the study eye (in eyes not included in the study IOP must have been controllable on no pharmacologic treatment or on the study medicine only)
* Best corrected visual acuity of 20/200 or better in the study eye(s)
* Ability of subject to understand character and individual consequences of clinical trial
* Signed and dated informed consent of the subject must be available before start of any specific trial procedures
* Women with childbearing potential have to practicing a medically accepted contraception during trial and a negative pregnancy test (serum or urine) should be existent before trial. Reliable contraception are systemic contraceptives (oral, implant, injection) and diaphragm or condoms with spermicidal. Women that are sterile by surgery or for more than two years postmenopausal can be participate in the trial.

Exclusion Criteria:

* Chronic or recurrent inflammatory eye disease
* Ocular trauma within the past six months
* Current ocular infection, i.e. conjunctivitis or keratitis
* Any abnormality preventing reliable applanation tonometry
* Intraocular surgery or laser treatment within the past three months
* Inability to discontinue contact lens wear during the study
* Use of any systemic medication that would affect IOP with less than a

  1-month stable dosing regimen before the screening visit
* Pregnancy and lactation
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product
* Participation in other clinical trials during the present clinical trial or within the last four weeks
* Medical or psychological condition that would not permit completion of the trial or signing of informed consent
* Subject is allergic to sulfonamides
* Severe renal dysfunction or hyperchloraemic acidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
intraocular pressure (IOP)-lowering | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Pfeiffer, Prof. Dr., Principal Investigator — Department of Opthalmology, Johannes Gutenberg University Mainz
Locations (1):
- Department of Opthalmology, Johannes-Gutenberg University Mainz, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Background] Hurvitz LM, Kaufman PL, Robin AL, Weinreb RN, Crawford K, Shaw B. New developments in the drug treatment of glaucoma. Drugs. 1991 Apr;41(4):514-32. doi: 10.2165/00003495-199141040-00002. PMID 1711957
- [Background] Distelhorst JS, Hughes GM. Open-angle glaucoma. Am Fam Physician. 2003 May 1;67(9):1937-44. PMID 12751655
- [Derived] Bell K, Korb C, Butsch C, Giers BC, Beck A, Strzalkowska A, Ruckes C, Klingberg U, Pfeiffer N, Lorenz K. A Randomized, Double-Masked, Active-Controlled, Crossover Phase III Equivalence Study of Generic Dorzolamide 2% versus Innovator Trusopt(R) Eye Drop Solution in Subjects with Open-Angle Glaucoma or Ocular Hypertension. J Ophthalmol. 2022 Jul 20;2022:5249922. doi: 10.1155/2022/5249922. eCollection 2022. PMID 35909461